CLINICAL TRIAL: NCT01595516
Title: Nebivolol and Endothelial Regulation of Fibrinolysis
Brief Title: Nebivolol and Endothelial Regulation of Fibrinolysis (NERF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Christopher DeSouza, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BYS-MD-72
Record Dates: First submitted 2012-03-05; First posted 2012-05-10 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Prehypertension; Hypertension
MeSH Terms: conditions — Prehypertension; Hypertension | interventions — Nebivolol; Metoprolol; Bradykinin; Sodium Chloride; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Nebivolol (Active Comparator)
  Interventions: Drug: Nebivolol
- Metoprolol (Active Comparator)
  Interventions: Drug: Metoprolol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Bradykinin (Other)
  Interventions: Drug: Nebivolol; Drug: Metoprolol; Drug: Placebo; Other: Bradykinin
- Saline (Other)
  Interventions: Drug: Nebivolol; Drug: Metoprolol; Drug: Placebo; Other: Bradykinin; Other: Saline; Other: Vitamin C
- Vitamin C (Other)
  Interventions: Drug: Nebivolol; Drug: Metoprolol; Other: Bradykinin; Other: Saline; Other: Vitamin C

INTERVENTIONS:
Drug: Nebivolol — 5 mg tablet to be taken by mouth once per day for 12 weeks
  Other Names: Bystolic
  Arms: Bradykinin; Nebivolol; Saline; Vitamin C
Drug: Metoprolol — 100 mg tablet to be taken by mouth once per day for 12 weeks
  Other Names: Toprol-XL
  Arms: Bradykinin; Metoprolol; Saline; Vitamin C
Drug: Placebo — Gelatin capsule to be taken by mouth once per day for 12 weeks
  Arms: Bradykinin; Placebo; Saline
Other: Bradykinin — Bradykinin is infused into the brachial artery at doses of 12.5, 25.0 and 50.0 ng/100 mL of forearm tissue /min. BDK stimulates the endothelial cells to release tissue type plasminogen activator (t-PA). Blood flow in mL/100 mL tissue/min is also measured to BDK.
  Other Names: BDK
  Arms: Bradykinin; Saline; Vitamin C
Other: Saline — Baseline or resting forearm blood flow is measured in response to saline for 5 minutes before each drug infusion. t-PA release in response to the saline is also measured.
  Arms: Saline; Vitamin C
Other: Vitamin C — The acute effects of into-arterial vitamin C on the ability of the endothelium to release t-PA was determined before and after the nebivolol and metoprolol intervention. After allowing sufficient time (~20 minutes) for FBF and plasma t-PA concentrations to return to baseline following the initial infusion of BDK, vitamin C (24 mg/min) was infused at a constant rate while the BDK dose-response curves were repeated. t-PA and FBF were measured.
  Arms: Saline; Vitamin C

SUMMARY:
The investigators hypothesize that nebivolol will improve endothelial t-PA release in adult humans with elevated blood pressure to a greater extent than either metoprolol or placebo. The investigators further hypothesize that the improvement in the capacity of the vascular endothelium to release t-PA with nebivolol is mediated, in part, by the compound's antioxidant properties.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be men and women of all races and ethnic backgrounds aged 45-65 years.
* Subjects will be prehypertensive/hypertensive defined as resting systolic blood pressure >125 mmHg and <160 mmHg and/or diastolic >80 mmHg and <100 mmHg.
* All of the women in the study will be postmenopausal and not receiving hormone replacement therapy (HRT) currently or in the preceding 3-year period.
* Candidates will be sedentary as determined from the Stanford Physical Activity Questionnaire (<35 kcal/wk) and will not have engaged in any program of regular physical activity for at least 1 year prior to the study.

Exclusion Criteria:

* Candidates who smoke (currently or in the past 7 years), report more than low-risk alcohol consumption as defined as no more than 14 standard drinks/wk and no more than 4 standard drinks/day for men and 7 standard drinks/wk and 3 standard drinks/day for women (a standard drink is defined as 12 ounces of beer, 5 ounces of wine, 1½ ounces of 80-proof distilled spirits).
* Potential candidates who are taking cardiovascular-acting (i.e. statins, blood pressure medication and aspirin) medications will not be eligible.
* Fasting plasma glucose >126 mg/dL.
* Potential candidates with a resting heart rate of < 50 beats/minute will be excluded.
* Use of hormone replacement therapy.
* In hypertensive subjects, a seated systolic blood pressure >160 mmHg or a seated diastolic blood pressure >100 mmHg will be excluded.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher DeSouza, Ph.D., Principal Investigator — University of Colorado at Boulder
Locations (1):
- UC-Boulder Clinical and Translational Research Center, Boulder, Colorado, United States

REFERENCES:
- [Derived] Stauffer BL, Dow CA, Diehl KJ, Bammert TD, Greiner JJ, DeSouza CA. Nebivolol, But Not Metoprolol, Treatment Improves Endothelial Fibrinolytic Capacity in Adults With Elevated Blood Pressure. J Am Heart Assoc. 2017 Nov 9;6(11):e007437. doi: 10.1161/JAHA.117.007437. PMID 29122812

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nebivolol | Metoprolol | Placebo
Started | 16 | 16 | 12
Completed | 16 | 16 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nebivolol | Metoprolol | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 12 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (5) | 58 (6) | 57 (6) | 58 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 16
  Male | 10 | 10 | 8 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 15 | 14 | 11 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 14 | 14 | 11 | 39
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 12 | 44

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate
Description: Resting heart rate in the seated position
Time Frame: Heart rate was measured before the 12 week drug or placebo intervention and after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Nebivolol | Metoprolol | Placebo
Number analyzed (Participants) | 16 | 16 | 12
bpm
  Before Intervention | 64 (1) | 71 (1) | 69 (2)
  After Intervention | 58 (2) | 64 (3) | 72 (2)

2. Primary Outcome: Systolic Blood Pressure
Time Frame: Systolic blood pressure was measured before the 12 week drug or placebo intervention and after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Nebivolol | Metoprolol | Placebo
Number analyzed (Participants) | 16 | 16 | 12
mmHg
  Before Intervention | 140 (2) | 138 (2) | 138 (2)
  After Intervention | 125 (2) | 125 (3) | 135 (3)

3. Primary Outcome: Diastolic Blood Pressure
Time Frame: Diastolic blood pressure was measured before the 12 week drug or placebo intervention and after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Nebivolol | Metoprolol | Placebo
Number analyzed (Participants) | 16 | 16 | 12
mmHg
  Before Intervention | 85 (2) | 87 (2) | 85 (3)
  After Intervention | 78 (2) | 79 (2) | 81 (2)

4. Primary Outcome: Endothelial t-PA Release in Response to Bradykinin (BDK) Before and After the 12 Week Intervention
Description: Net endothelial release of t-PA antigen in response to bradykinin (BDK) was calculated using the following equation: Net Release of t-PA Antigen=(Cv-Ca) x (FBF x [101-hematocrit/100]) where Cv and Ca represent the concentration of t-PA in the vein and artery respectively. A positive difference indicates a net release and a negative difference net uptake. Arterial and venous blood samples are collected simultaneously at baseline and each dose of the drug (BDK). t-PA concentration were determined by enzyme immunoassay. Hematocrit was measured in triplicate using the standard microhematocrit technique and corrected for trapped plasma volume within the trapped red blood cells.
Time Frame: t-PA release was measured before the 12 week drug or placebo intervention and after the 12 week drug or placebo intervention.
Measure: Mean (Standard Error); unit: ng/100 mL tissue/min
Groups:
- Before Nebivolol: Before randomization to nebivolol
- After Nebivolol: Nebivolol: 5 mg tablet to be taken by mouth once per day for 12 weeks
- Before Metoprolol: Before randomization to metoprolol
- After Metoprolol: Metoprolol: 100 mg tablet to be taken by mouth once per day for 12 weeks
- Before Placebo: Before randomization to placebo
- After Placebo: Placebo: Gelatin capsule to be taken by mouth once per day for 12 weeks
Arm/Group | Before Nebivolol | After Nebivolol | Before Metoprolol | After Metoprolol | Before Placebo | After Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 12 | 12
ng/100 mL tissue/min
  Amount of t-PA release to Saline | -1.2 (0.8) | -1.8 (0.9) | -1.2 (1.2) | -1.9 (1.1) | -0.2 (1.2) | -0.9 (1.5)
  Amount of t-PA release to BDK 12.5 | 15.7 (2.9) | 25.2 (4.1) | 14.4 (3.3) | 16.6 (3.3) | 18.1 (3.1) | 17.6 (2.8)
  Amount of t-PA release to BDK 25.0 | 29.1 (3.9) | 46.4 (6.5) | 27.5 (3.3) | 31.2 (2.4) | 28.3 (3.8) | 32.7 (5.6)
  Amount of t-PA release to BDK 50.0 | 47.2 (4.3) | 72.8 (5.7) | 48.2 (5.9) | 52.7 (4.6) | 51.1 (5.0) | 52.9 (4.3)

5. Primary Outcome: Endothelial t-PA Release in Response to Bradykinin (BDK) and Bradykinin+Vitamin C (BDK+C) Before and After 12 Weeks of Nebivolol Therapy.
Description: Net endothelial release of t-PA antigen in response to bradykinin (BDK) and bradykinin+vitamin C (BDK+C) was calculated using the following equation: Net Release of t-PA Antigen=(Cv-Ca) x (FBF x [101-hematocrit/100]) where Cv and Ca represent the concentration of t-PA in the vein and artery respectively. A positive difference indicates a net release and a negative difference net uptake. Arterial and venous blood samples are collected simultaneously at baseline and each dose of the drug (BDK) and BDK+Vit C. t-PA concentration were determined by enzyme immunoassay. Hematocrit was measured in triplicate using the standard microhematocrit technique and corrected for trapped plasma volume within the trapped red blood cells.
Time Frame: t-PA release was measured before the 12 week drug intervention and after the 12 week drug intervention.
Measure: Mean (Standard Error); unit: ng/100 mL tissue/min
Groups:
- Before Nebivolol: Saline: Net t-PA antigen release in response to BDK before 12 weeks of nebivolol therapy.
- Before Nebivolol: Vitamin C: Net t-PA antigen release in response to BDK+C before 12 weeks of nebivolol therapy.
- After Nebivolol: Saline: Net t-PA antigen release in response to BDK after 12 weeks of nebivolol therapy.
- After Nebivolol: Vitamin C: Net t-PA antigen release in response to BDK+C after 12 weeks of nebivolol therapy.
Arm/Group | Before Nebivolol: Saline | Before Nebivolol: Vitamin C | After Nebivolol: Saline | After Nebivolol: Vitamin C
Number analyzed (Participants) | 10 | 10 | 10 | 10
ng/100 mL tissue/min
  Amount of t-PA release to saline | -2.4 (1.1) | -1.4 (0.8) | -1.5 (1.3) | -3.8 (2.6)
  Amount of t-PA release to BDK 12.5 | 14.3 (3.2) | 31.3 (5.5) | 28.2 (6.2) | 38.1 (7.3)
  Amount of t-PA release to BDK 25.0 | 27.6 (5.0) | 52.7 (6.6) | 49.1 (9.1) | 54.2 (7.9)
  Amount of t-PA release to BDK 50.0 | 47.2 (5.0) | 80.5 (6.2) | 67.5 (7.1) | 79.9 (7.6)

6. Primary Outcome: Endothelial t-PA Release in Response to BDK and BDK+C Before and After 12 Weeks of Metoprolol Therapy.
Description: Net endothelial release of t-PA antigen in response to BDK and BDK+C was calculated using the following equation: Net Release of t-PA Antigen=(Cv-Ca) x (FBF x [101-hematocrit/100]) where Cv and Ca represent the concentration of t-PA in the vein and artery respectively. A positive difference indicates a net release and a negative difference net uptake. Arterial and venous blood samples are collected simultaneously at baseline and each dose of the drug (BDK) and BDK+Vit C. t-PA concentration were determined by enzyme immunoassay. Hematocrit was measured in triplicate using the standard microhematocrit technique and corrected for trapped plasma volume within the trapped red blood cells.
Time Frame: t-PA release was measured before the 12 week drug intervention and after the 12 week drug intervention.
Measure: Mean (Standard Error); unit: ng/100 mL tissue/min
Groups:
- Before Metoprolol: Saline: Net t-PA antigen release in response to BDK before 12 weeks of nebivolol therapy.
- Before Metoprolol: Vitamin C: Net t-PA antigen release in response to BDK+C before 12 weeks of nebivolol therapy.
- After Metoprolol: Saline: Net t-PA antigen release in response to BDK after 12 weeks of nebivolol therapy.
- After Metoprolol: Vitamin C: Net t-PA antigen release in response to BDK+C after 12 weeks of nebivolol therapy.
Arm/Group | Before Metoprolol: Saline | Before Metoprolol: Vitamin C | After Metoprolol: Saline | After Metoprolol: Vitamin C
Number analyzed (Participants) | 10 | 10 | 10 | 10
ng/100 mL tissue/min
  Amount of t-PA release to Saline | -2.7 (0.9) | -2.5 (0.8) | -1.3 (1.4) | -2.7 (1.1)
  Amount of t-PA release to BDK 12.5 | 10.1 (3.9) | 31.1 (5.0) | 16.4 (5.0) | 30.0 (4.4)
  Amount of t-PA release to BDK 25.0 | 24.5 (3.8) | 47.1 (7.3) | 31.3 (3.3) | 46.4 (6.3)
  Amount of t-PA release to BDK 50.0 | 45.0 (5.5) | 82.4 (10.2) | 49.9 (5.7) | 73.8 (7.4)

ADVERSE EVENTS:
Time Frame: Adverse event data for each participant was assessed every 2 weeks during their check-in visits at the CU-Boulder CTRC over the 12 weeks.
Arm/Group | Nebivolol | Metoprolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT01595516/Prot_SAP_000.pdf